CLINICAL TRIAL: NCT06835166
Title: Effect of Intraoperative Position Change on Hemodynamics and Cardiac Electrophysiological Balance Index in Morbidly Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy
Brief Title: Effect of Intraoperative Position Change on Hemodynamics and Electrocardiography
Status: Completed | Type: Observational
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Fatma Çelik, Assoc. Prof. Dr., Firat University
Other Study IDs: FiratU-ANEST-FC-01
Record Dates: First submitted 2025-02-06; First posted 2025-02-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Bariatric Surgery (Sleeve Gastrectomy ); Hemodynamics; Electrocardiography
Keywords: Bariatric Surgery; Laparoscopic sleeve gastrectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: 12-lead electrocardiography measurement — Intraoperative 12-lead electrocardiography (EKG) measurement during laparoscopic sleeve gastrectomy in morbidly obese patients:
  In all patients, pneumoperitoneum CO₂ intraabdominal pressure will be studied as 15 cmH₂O.
  Intraoperatively, 12-lead ECG will be obtained at five position measurement points:
  Procedure1. Supine-monitored; Procedure 2. After induction; Procedure 3. Under general anesthesia-Supine-abdominal inflated; Procedure 4. Abdominal inflated-(30% vertical) Reverse Trendelenburg; Procedure 5. Abdominal deflated-(30% vertical) Reverse Trendelenburg.
  Hemodynamic monitoring [systolic blood pressure, diastolic blood pressure, mean arterial pressure, heart rate ] was recorded at 5 simultaneous measurement points.
  All hemodynamic measurements and ECG recordings will be performed 3 minutes after the position change to ensure standardization, to allow the response to settle after the position change, and to prevent the possibility of exaggerated-incorrect data.

SUMMARY:
The combined effects of obesity-related cardiac structure and function changes, comorbidities, pneumoperitoneum technique, and reverse Trendelenburg position may complicate anesthesia management by affecting intraoperative hemodynamics and cardiac function. Increased intra-abdominal pressure leads to various physiological changes through mechanical and neurohormonal responses. Furthermore, pneumoperitoneum and reverse Trendelenburg position are reported to stimulate the sympathetic nervous system and increase the risk of cardiac arrhythmia.

Obesity-related changes in cardiac structure and function have been shown to predispose to cardiac conduction and repolarization disorders. It has also been stated that obesity directly affects cardiac electrophysiology.

Moreover, obese patients may have hidden risks associated with the development of cardiac arrhythmias due to the adverse contributions of the cardiovascular effects of anesthesia, pneumoperitoneum, and patient positioning during laparoscopic intervention.

The index of cardiac electrophysiological balance (iCEB) is a non-invasive marker calculated by the QT/QRS ratio that can predict malignant ventricular arrhythmias.

The aim of this study was to investigate the effects of intraoperative patient positions on hemodynamics and the index of cardiac electrophysiological balance (iCEB) during laparoscopic sleeve gastrectomy in morbidly obese patients.

DETAILED DESCRIPTION:
Morbidly obese patients who will undergo laparoscopic sleeve gastrectomy will be included in the study.

Patients will be taken to the operating room without premedication after a minimum of 8 hours of fasting. Venous access will be established with a 22 G angiocatheter on the operating table. Routine heart rate, arterial blood pressure, peripheral oxygen saturation (SpO₂), body temperature, bispectral index (BIS) (Bispectral Drager Vista 120 system, Covidien, USA) monitoring will be performed. BIS will be kept between 40 - 60. In addition, 12-lead ECG (Cardioline®) will be used for electrocardiogram (ECG) measurements.

Mechanical ventilation will be provided with a tidal volume of 8 mL/kg (IBW) and a positive end expiratory pressure (PEEP) of 8 cmH₂O. The respiratory rate will be adjusted to maintain end-tidal carbon dioxide (EtCO2) at 35 to 45 mmHg.

Targeted Fluid Management (GDFM) will be provided by continuous Pleth Variability Index (PVI) monitoring by placing a Pulse CO-Oximeter sensor system (Masimo rainbow set® Masimo Corporation, Irvine, CA, USA) on the patients' 4th finger. Hemodynamic targets are both PVI and mean arterial pressure. Fluid loading prescription is based on a PVI value greater than 13%, and vasopressor use is based on a mean arterial pressure < 65 mmHg. If necessary, additional fluids and norepinephrine will be given to maintain mean arterial pressure > 65 mmHg.

A 12-lead ECG will be taken at five intraoperative position measurement points (1. Supine-monitored; 2. After induction; 3. Under general anesthesia-Supine-abdominal inflated; 4. Abdominal inflated-(30% upright) Reverse Trendelenburg; 5. Abdominal deflated-(30% upright) Reverse Trendelenburg). Hemodynamic monitoring [systolic blood pressure (SBP), diastolic blood pressure (DAB), mean arterial pressure (MAP), heart rate (HR)] will be recorded at 5 simultaneous measurement points. All hemodynamic measurements and ECG recordings will be made 3 minutes after the position change to ensure standardization, allow the response to settle after the position change, and prevent the possibility of exaggerated or false data.

All patients will have their surgeries performed by the same surgical team and intra-abdominal pressure will be kept below 15 mmHg.

Demographic data (age, gender, height, weight, BMI), American Society of Anesthesiologists (ASA) physical status classification, preoperative assessment information (comorbidities, medications used), duration of surgery and anesthesia, amount of fluid administered, and amount of norepinephrine to be used when needed will be recorded.

Power analysis was calculated as follows:

Repeated measures, within factors Options: Pillai V, O'Brien-Shieh Algorithm Analysis: A priori: Compute required sample size Input: Effect size f = 0.25 α = 0.05 Power (1-β ) = 0.95 Number of groups = 1 Number of measurements = 5 Corr among rep measures = 0 Output: Noncentrality parameter λ = 20.3125000 Critical F = 2.5226149 Numerator df = 4.0000000 Denominator df = 61.0000000 Total sample size = 65 Actual power = 0.9523977 Pillai V = 0.2380952 Considering that there may be data loss in ECG measurements and evaluations, the number of cases was determined as 80 patients.

Intraoperative hemodynamic and ECG (Heart-electrophysiological balance index (iCEB = QT/QRS ratio) changes in 5 positions will be evaluated.

ELIGIBILITY:
Inclusion criteria:

1. Adult patient planned for elective primary laparoscopic sleeve gastrectomy surgery
2. Body Mass Index (BMI) ≥ 40 kg/ / m²
3. Age ≥ 18
4. ASA physical health class II-III.

Exclusion criteria:

1. Patient refusal to participate in the study
2. Those who underwent revision laparoscopic sleeve gastrectomy
3. Emergency laparoscopic sleeve gastrectomy surgery (stump leakage, etc.)
4. Secondary surgery in addition to elective laparoscopic sleeve gastrectomy
5. Patients with previous recurrent abdominal surgery
6. Patients with electrolyte imbalance
7. Direct laryngoscopy in ramp position
8. Multiple intubation attempts due to difficult intubation
9. Preoperative arrhythmia and heart failure (ejection fraction < 30%)
10. Renal and liver failure
11. Patients who require > 8 ml/kg for tidal volume

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbidly obese patients undergoing laparoscopic sleeve gastrectomy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of the QT (ms) interval in morbidly obese patients undergoing laparoscopic sleeve gastrectomy. | The operation takes approximately 2 hours to complete.
  Electrocardiograms will be recorded in the following predefined positions:
  1. Supine - monitored; 2. Post-anesthesia; 3. Under general anesthesia - Supine - abdominal distension; 4. Abdominal distension - (30% vertical) Reverse Trendelenburg; 5. Abdominal distension reduced - (30% vertical) Reverse Trendelenburg)
Evaluation of QRS (ms) interval in morbidly obese patients undergoing laparoscopic sleeve gastrectomy. | The operation takes approximately 2 hours to complete.
  Electrocardiograms will be recorded in the following predefined positions:
  (1. Supine - monitored; 2. Post-anesthesia; 3. Under general anesthesia - Supine - abdominal distension; 4. Abdominal distension - (30% vertical) Reverse Trendelenburg; 5. Abdominal distension reduced - (30% vertical) Reverse Trendelenburg)
Evaluation of the cardiac electrophysiological balance index (QT/QRS) in morbidly obese patients undergoing laparoscopic sleeve gastrectomy. | The operation takes approximately 2 hours to complete.
  The QT interval will be measured from the beginning of the QRS complex to the end of the T wave, and the QT/QRS (iCEB) ratio will be calculated.
Patient height measurement (in meters) | Height measurement for each patient takes approximately 10 minutes.
  All patients' heights will be measured (in meters).
Patients' body weight measurement (kilograms) | Body weight measurement takes approximately 10 minutes for each patient.
  Patients' body weights will also be measured (in kilograms).
Calculation of body mass index (BMI = kg/m²). | This will take approximately 10 minutes for each patient.
  Body Mass Index (BMI) is calculated by dividing body weight (kg) by the square of height (m) (BMI = kg/m²).

SECONDARY OUTCOMES:
Evaluation of patients' blood pressure measurements (mmHg) | The operation takes approximately 2 hours to complete.
  Patients' blood pressure will be recorded as systolic, diastolic, and mean blood pressure.
  Measurement time points are indicated below:
  (1. Supine - monitored; 2. Post-anesthesia; 3. Under general anesthesia - Supine - abdominal distension; 4. Abdominal distension - (30% vertical) Reverse Trendelenburg; 5. Abdominal distension reduced - (30% vertical) Reverse Trendelenburg)
measurement of patients' heart rates (beats/min) | The operation takes approximately 2 hours to complete.
  Measurement time points are indicated below:
  (1. Supine - monitored; 2. Post-anesthesia; 3. Under general anesthesia - Supine - abdominal distension; 4. Abdominal distension - (30% vertical) Reverse Trendelenburg; 5. Abdominal distension reduced - (30% vertical) Reverse Trendelenburg)

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Çelik, Assoc. Dr., Principal Investigator — fatma.celik@firat.edu.tr
Locations (1):
- Firat University Hospital, Department of Anesthesiology and Reanimation, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We have not yet decided whether to share the IPDs of our study.

REFERENCES:
- [Background] Atkinson TM, Giraud GD, Togioka BM, Jones DB, Cigarroa JE. Cardiovascular and Ventilatory Consequences of Laparoscopic Surgery. Circulation. 2017 Feb 14;135(7):700-710. doi: 10.1161/CIRCULATIONAHA.116.023262. PMID 28193800
- See also: Echocardiographic and hemodynamic evaluation of cardiovascular performance during laparoscopy of morbidly obese patients — https://pubmed.ncbi.nlm.nih.gov/14627473/
- See also: Evaluation of index of cardio-electrophysiological balance in patients with coronary slow flow — https://pubmed.ncbi.nlm.nih.gov/34218730/